CLINICAL TRIAL: NCT03228290
Title: Functional Assessment in Liver Transplant Candidates (FrAILT) Study
Brief Title: Functional Assessment in Liver Transplantation
Acronym: FrAILT
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11-07513; 1R21AG067554 (NIH); R21DK127275 (NIH)
Record Dates: First submitted 2017-05-04; First posted 2017-07-24 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: End Stage Liver Disease
Keywords: Cirrhosis; Liver; Liver Transplant; Frailty; end stage
MeSH Terms: conditions — End Stage Liver Disease; Fibrosis; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sub-group of 1000 patients will have one single blood draw of 2 tablespoons of blood and provide a urine and stool sample (about 5ml each or 1 teaspoon each), at the time of consent. If they agree to participate in the DNA genetic testing, then they will have an additional 1 tablespoon drawn during the same venipuncture.
  Sub-group of 1000 patients will have adipose, muscle, liver tissue, and blood collected during the liver transplant surgery.
  * 8 cm³ of muscle tissue from the rectus muscle in the abdomen.
  * 8 cm³ of adipose tissue from the subcutaneous and visceral adipose tissue of the abdomen.
  * 8 cm³ of liver tissue from the explanted liver
  * 4 tablespoons of blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This will be a prospective cohort study of patients with liver disease. Subjects will undergo geriatric assessments of frailty, functional status, and disability using functional status measures at baseline and at every clinic visit in the pre-transplant setting. Subjects will also answer questions regarding quality of life, personality, and/or cognitive function. Subjects will again undergo assessments at every clinic visit through 12 months after transplant. Then, they will be followed annually.

DETAILED DESCRIPTION:
Patients will be asked to perform the following study procedures:

1. Assessment of cognitive function, quality of life, and/or personality using cognitive tests and questionnaires.
2. Measures of frailty and disability selected to capture the multi-dimensional aspects of frailty including functional status and physiologic reserve:

   Fried Frailty Score: weakness (test of grip strength), exhaustion (patient interview), slowness (gait speed), low activity (patient interview) Short Physical Performance Battery: repeated chair stands, balance testing with feet together, 13-foot walk
3. Laboratory tests will all be obtained from the medical record: creatinine, total bilirubin, INR, sodium, albumin. All of these tests are necessary for listing for liver transplantation.
4. Blood draw, urine and stool samples will be collected for a sub-group of 1000 patients.
5. Adipose, muscle, liver tissue, and blood will be collected during the liver transplant surgery for a sub-group of 1000 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* Are seen for the treatment of liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are being seen for the treatment of their liver disease.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2011-10-12 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Frailty and functional status as assessed by grip strength, chair stands, and balance which comprise the Liver Frailty Index (LFI). | December 31, 2023
  Grip strength: Performance-based. Measured in kilograms. This was measured in each subject's dominant hand using a hand dynamometer (Jamar Hydraulic hand dynamometer). We averaged three trials.
  Chair stands: Performance-based. Measured in number of chair stands per second. Number of chair stands completed in 30 seconds.
  Balance: Performance-based. Measured in seconds. Ability to balance in three positions (feet placed side to side, semitandem, and tandem) for 10 seconds each.
  Liver Frailty Index (LFI): (coefficient x grip) + (coefficient x chair stands) + (coefficient x balance) +6
Examine the association between frailty and outcomes both before and after liver transplantation. | December 31, 2023
  Outcomes measured prior to transplant will include: waiting for transplant, died pre-transplant, deactivated too sick, deactivated for social reasons/inactive, deferred not a candidate, and transplanted. Outcomes that will be measured post transplant include: still alive, died post transplant, and re-transplanted. All measures will be acquired via patient interview or review of medical records.
Evaluate the change in frailty and physical function both before and after liver transplant or treatment utilizing the LFI. | December 31, 2023
  See outcome 1 for how LFI is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Lai, MD, MBA, Principal Investigator — University of California, San Francisco
Locations (12):
- United States (12):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Loma Linda University, Loma Linda, California
  - University of California, San Francisco, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor Scott & White Health, Dallas, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lai JC, Feng S, Terrault NA, Lizaola B, Hayssen H, Covinsky K. Frailty predicts waitlist mortality in liver transplant candidates. Am J Transplant. 2014 Aug;14(8):1870-9. doi: 10.1111/ajt.12762. Epub 2014 Jun 16. PMID 24935609
- [Result] Lai JC, Covinsky KE, Hayssen H, Lizaola B, Dodge JL, Roberts JP, Terrault NA, Feng S. Clinician assessments of health status predict mortality in patients with end-stage liver disease awaiting liver transplantation. Liver Int. 2015 Sep;35(9):2167-73. doi: 10.1111/liv.12792. Epub 2015 Feb 12. PMID 25644788
- [Result] Wang CW, Covinsky KE, Feng S, Hayssen H, Segev DL, Lai JC. Functional impairment in older liver transplantation candidates: From the functional assessment in liver transplantation study. Liver Transpl. 2015 Dec;21(12):1465-70. doi: 10.1002/lt.24334. Epub 2015 Nov 6. PMID 26359787
- [Result] Lai JC, Dodge JL, Sen S, Covinsky K, Feng S. Functional decline in patients with cirrhosis awaiting liver transplantation: Results from the functional assessment in liver transplantation (FrAILT) study. Hepatology. 2016 Feb;63(2):574-80. doi: 10.1002/hep.28316. Epub 2015 Dec 16. PMID 26517301
- [Result] Wang CW, Feng S, Covinsky KE, Hayssen H, Zhou LQ, Yeh BM, Lai JC. A Comparison of Muscle Function, Mass, and Quality in Liver Transplant Candidates: Results From the Functional Assessment in Liver Transplantation Study. Transplantation. 2016 Aug;100(8):1692-8. doi: 10.1097/TP.0000000000001232. PMID 27314169
- [Result] Lai JC, Volk ML, Strasburg D, Alexander N. Performance-Based Measures Associate With Frailty in Patients With End-Stage Liver Disease. Transplantation. 2016 Dec;100(12):2656-2660. doi: 10.1097/TP.0000000000001433. PMID 27495749
- [Result] Sinclair M, Poltavskiy E, Dodge JL, Lai JC. Frailty is independently associated with increased hospitalisation days in patients on the liver transplant waitlist. World J Gastroenterol. 2017 Feb 7;23(5):899-905. doi: 10.3748/wjg.v23.i5.899. PMID 28223735
- [Derived] Berry KA, Kent D, Seetharaman S, Wong R, Mohamad Y, Yao F, Nunez-Duarte M, Wadhwani SI, Boyarsky BJ, Rahimi RS, Duarte-Rojo A, Kappus MR, Volk ML, Ladner DP, Segev DL, McAdams-DeMarco M, Verna EC, Ganger DR, Lai JC. Loneliness in adults awaiting liver transplantation at 7 U.S. transplant centers. Ann Hepatol. 2022 Sep-Oct;27(5):100718. doi: 10.1016/j.aohep.2022.100718. Epub 2022 Apr 20. PMID 35460882
- [Derived] Berry K, Duarte-Rojo A, Grab JD, Dunn MA, Boyarsky BJ, Verna EC, Kappus MR, Volk ML, McAdams-DeMarco M, Segev DL, Ganger DR, Ladner DP, Shui A, Tincopa MA, Rahimi RS, Lai JC; from the Multi-Center Functional Assessment in Liver Transplantation (FrAILT) Study. Cognitive Impairment and Physical Frailty in Patients With Cirrhosis. Hepatol Commun. 2022 Jan;6(1):237-246. doi: 10.1002/hep4.1796. Epub 2021 Aug 24. PMID 34558844
- See also: We developed a novel clinical liver frailty index, consisting of hand grip strength, timed chair stands, and balance testing, that correctly reclassifies 1 in 5 patients to their accurate survival status, compared to MELDNa alone. — http://liverfrailtyindex.ucsf.edu/